CLINICAL TRIAL: NCT00200265
Title: Changing Eating Behaviors in Young Children: Should Healthy Foods be Increased or Unhealthy Foods Decreased?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7-05-HFC-27
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2007-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet

ARMS (3):
- 1 (Experimental): Behavioral: diet
  Interventions: Behavioral: diet
- 2 (Experimental): Behavioral: diet
  Interventions: Behavioral: diet
- 3 (Placebo Comparator): Behavioral: diet
  Interventions: Behavioral: diet

INTERVENTIONS:
Behavioral: diet — diet

SUMMARY:
Recommendations for treatment of childhood obesity in a primary care setting have been developed. These recommendations include beginning treatment with young children, focusing treatment on the parent so the parent can assist the child in making changes, and changing 2 or 3 very specific eating or activity behaviors (i.e., eat less snacks, rather than eat less calories). The effectiveness of these recommendations has never been evaluated. This project's goal is to develop, implement, and evaluate a 6-month childhood obesity intervention meeting these recommendations. Another goal of the project is to compare two different approaches, focusing on either decreasing intake of two unhealthy foods or increasing intake of two healthy foods, for changing eating behaviors during treatment. Two hundred ten children, between the ages of 4 to 9 years, who are at risk for overweight or overweight, based upon weight and height standards, will be randomized to one of three treatments: 1) a Newsletter treatment (provided with information on healthy eating only); 2) a Parent Program that decreases intake of sweet/salty snack foods (< 3 servings/week) and sweetened drinks (< 3 servings/week); or 3) a Parent Program that increases intake of fruits and vegetables (5 servings/day) and low-fat dairy products (2 servings/day). Children's height and weight will be measured at 0, 3, 6, 9, and 12 months. This project will determine if the recommendations for treatment are effective, and if focusing on decreasing intake of unhealthy foods or increasing intake of healthy foods produces a better long-term weight loss outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 4 and 9 years. We propose to use this age group since parents are in control of the eating and exercise choices of such children, and thus a program that focuses on parenting behaviors (i.e., positive reinforcement, stimulus control, parental modeling) should be developmentally appropriate. This age group also meets the Expert Committee's goal of intervening early5; moreover children aged 4 to 8 years have similar nutritional needs.
2. Body mass index (BMI) > 85th percentile BMI. Based upon the Expert Committee recommendations,5 children > 2 years of age who are identified as being at risk for overweight (85th to 94th percentile BMI) or overweight (> 95th percentile BMI) should focus on weight maintenance as height continues to increase. These recommendations are aimed at reducing z-BMI.
3. Tanner stage 1 (prepubertal) sexual maturation status.
4. Self-report at least one of the following problematic behaviors:

   1. Consume < 2 servings per day of whole fruit (not juice) or < 3 servings per day of vegetables.
   2. Consume > 1 serving of sweetened drink per day.
   3. Consume < 2 servings of low-fat milk per day.
   4. Consume > 4 times per week of sweet or salty snack foods.
5. A parent willing to attend treatment meetings.
6. Parent and child speak English.

   -

Exclusion Criteria:

1. Report a family member participating in another weight loss program.
2. Report that the child or parent planning to attend the treatment meetings has a major psychiatric disease or organic brain syndrome.
3. Report that the child or parent planning to attend the treatment meetings has dietary or physical activity restrictions.
4. Intend to move outside of the metropolitan area within the time frame of the investigation.

   -

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2005-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
z-BMI in children | 12 months

SECONDARY OUTCOMES:
Eating and activity behaviors | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Hart CN, Raynor HA, Osterholt KM, Jelalian E, Wing RR. Eating and activity habits of overweight children on weekdays and weekends. Int J Pediatr Obes. 2011 Oct;6(5-6):467-72. doi: 10.3109/17477166.2011.590204. Epub 2011 Jul 20. PMID 21774578
- [Derived] Raynor HA, Osterholt KM, Hart CN, Jelalian E, Vivier P, Wing RR. Evaluation of active and passive recruitment methods used in randomized controlled trials targeting pediatric obesity. Int J Pediatr Obes. 2009;4(4):224-32. doi: 10.3109/17477160802596189. PMID 19922036